CLINICAL TRIAL: NCT04151875
Title: Effect of Extraction Versus Non-extraction Orthodontic Treatment on Vertical Facial Dimension: A Non-Randomized Clinical Trial
Brief Title: Effect of Extraction Vs Non-extraction Orthodontic Treatment on Vertical Facial Dimension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hasan Abdullah Naji Hasan, Principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTH 3-3-4 CU
Record Dates: First submitted 2019-10-18; First posted 2019-11-05 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Malocclusion; Long Face Syndrome; Crowding, Tooth
Keywords: orthodontics; vertical dimension; premolars extraction; long face
MeSH Terms: conditions — Malocclusion | interventions — Braces; Tooth Extraction

STUDY DESIGN:
Intervention Model Description: -Interventions Intervention Group (I) Extraction treatment group. Bonding all cases will be performed by the principal investigator, then premolars extraction will be done, then installing the 1st alignment wire.
  Comparator group (C):
  Non-extraction group. Same orthodontist will bond all the cases and install the 1st alignment wire.
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor will be masked about the group of the participant during the measuring the outcome ..
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extraction orthodontic treatment (Experimental): orthodontic treatment with teeth extraction
  Interventions: Device: Extraction orthodontic treatment
- Non-extraction orthodontic treatment (Active Comparator): non-extraction orthodontic treatment
  Interventions: Device: Non-extraction orthodontic treatment

INTERVENTIONS:
Device: Extraction orthodontic treatment — orthodontic treatment with teeth extraction
  Other Names: Braces with teeth extraction
  Arms: Extraction orthodontic treatment
Device: Non-extraction orthodontic treatment — Non-extraction orthodontic treatment
  Other Names: Braces with no extraction of teeth
  Arms: Non-extraction orthodontic treatment

SUMMARY:
The aim of the current clinical trial was to evaluate the effects of premolar extractions compared with non-extraction orthodontic treatment on the skeletal vertical dimension of the face.

The null-hypothesis is that there is no difference in post-treatment skeletal vertical characteristics of normodivergent and hyperdivergent patients treated orthodontically with first premolar extractions compared with patients treated in non-extraction manner.

DETAILED DESCRIPTION:
The current protocol will be submitted for partial fulfillment of the PhD requirements in Faculty of Dentistry, Cairo University.

The trial will be conducted in the outpatient clinic of the Orthodontic Department, Faculty of Dentistry, Cairo University.

Primary examination and diagnosis of the patients seeking orthodontic treatment will be performed, to select a sample of the trial.

then, final diagnosis and planing of each participant will be performed by a trained orthodontists to be sure that all patients fallen with the inclusion criteria.

Interventions will be conducted with the same orthodontist, under supervision of orthodontic professors in the Orthodontic department, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* Normodivergent and hyperdivergent patients
* Cases with moderate crowding.
* Borderline cases which could be treated with extraction or non-extraction strategies

Exclusion Criteria:

* Hypodivergent patients.
* Cases with extremely sever crowding.
* Patients with high caries index or periodontal problems.
* Patients with systemic diseases, or syndromic conditions.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Vertical Dimension (VD) | after 1year. Changes will be measured before the start of trial and at the end of space closing stage, which anticipated to be within 12 months of intervention
  Vertical dimension of the face will be assessed by measuring a distances in millimeters between vertical points as ANS-Me (lower facial height), also it will be measured form angles in a degrees as angle SN/MP

SECONDARY OUTCOMES:
Changes in Overbite | 1 year . Changes will be measured before the start of trial and at the end of space closing stage, which anticipated to be within 12 months of intervention
  Distances in millimeters will be measure directly in patient mouth by using caliper it will be measured in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan A Alrubaie, MSc, Principal Investigator — Orthodontic department, Faculty of Dentistry, Cairo University; Amira A Aboulnaga, PhD, Study Director — Orthodontic department, Faculty of Dentistry, Cairo University; Mai H Aboulfotouh, PhD, Study Director — Orthodontic department, Faculty of Dentistry, Cairo University; Amr E El dakroury, Prof., Study Chair — Orthodontic department, Faculty of Dentistry, Cairo University
Locations (1):
- Hasan Hasan, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
it will be shareable for any researcher
Supporting Information: Study Protocol
Time Frame: within month it will be ready
Access Criteria: no special criteria..any orthodontic researcher can access the data

REFERENCES:
- [Derived] Alrubaie HA, Aboalnaga AA, Alhammadi MS, Eldakroury AE, Aboulfotouh MH. Vertical skeletal dimension and dentoalveolar changes in extraction versus non-extraction orthodontic treatment in class I malocclusion: a non-randomized clinical trial. Clin Oral Investig. 2026 Feb 4;30(2):69. doi: 10.1007/s00784-026-06768-0. PMID 41636882